CLINICAL TRIAL: NCT03583554
Title: Electrophysiological Biomarkers of Kynurenine Pathway Modulator AV-101 in Healthy Volunteers: Treating Suicidal Veterans
Brief Title: Electrophysiological Biomarkers of AV-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Marijn Lijffijt, PhD (Other)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency); VistaGen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Marijn Lijffijt, PhD, Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-41830
Record Dates: First submitted 2018-05-16; First posted 2018-07-11 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: Suicide; Kynurenine; metabolic pathway; Veterans; OEF/OIF/OND; electrophysiology; NMDA receptor; suicidal ideation
MeSH Terms: conditions — Suicide; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: placebo-controlled, randomized, double-blind, cross-over
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The research pharmacist compiles and has unique access to the randomization key
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo, then AV-101 720mg, then AV-101 1440mg (Placebo Comparator): Participants first received oral placebo. After at least 3 days wash-out participants get oral AV-101 720mg (matching placebo capsules). After at least 3 days wash-out participants get oral AV-101 1440mg (matching placebo capsules).
  Interventions: Drug: Placebo; Drug: AV-101 720 mg; Drug: AV-101 1440 mg
- AV-101 720mg, then AV-101 1440mg, then placebo (Experimental): Participants first received oral AV-101 720mg (matching placebo capsules). After at least 3 days wash-out participants get oral AV-101 1440mg (matching placebo capsules). After at least 3 days wash-out participants get oral placebo.
  Interventions: Drug: Placebo; Drug: AV-101 720 mg; Drug: AV-101 1440 mg
- AV-101 1440mg, then placebo, then AV-101 720mg (Experimental): Participants first received oral AV-101 1440mg (matching placebo capsules). After at least 3 days wash-out participants get oral placebo. After at least 3 days wash-out participants get oral AV-101 720mg (matching placebo capsules).
  Interventions: Drug: Placebo; Drug: AV-101 720 mg; Drug: AV-101 1440 mg

INTERVENTIONS:
Drug: Placebo — Single dose of 4 placebo oral capsules
  Other Names: Placebo oral dose
Drug: AV-101 720 mg — Single dose of 2 360 mg AV-101 oral capsules + 2 placebo oral capsules
  Other Names: L-4-Chlorokynurenine
Drug: AV-101 1440 mg — Single dose of 4 360 mg AV-101 oral capsules
  Other Names: L-4-Chlorokynurenine

SUMMARY:
Suicide is 2-7x higher in Veterans than non-veterans, and may be related to brain kynurenine pathway (KP) dysregulation and NMDA receptor (NMDAR) hyperactivation. Experimental drug "AV-101" modulates the brain KP, with possible downstream NMDAR deactivation. The investigators will examine AV-101 NMDAR modulation by testing dose-response effects on resting state EEG, Mismatch Negativity, and P50 gating. Twelve healthy Operation Enduring Freedom (OEF) Operation Iraqi Freedom (OIF) and Operation New Dawn (OND) Veterans will be administered single dose AV-101 720 mg, 1440 mg, and placebo over 3 weeks in a randomized, double-blind, cross-over trial. Repeated measures General Linear Models will test dose-response effects. Suicide prevention is an important Veterans Affair (VA) mission. This study is a first step to testing anti-suicidal effects of AV-101 in Veterans.

DETAILED DESCRIPTION:
Background: Suicide is the 10th leading cause of death in the US, and is 2-7 times higher in Veterans than age- and sex-matched civilians. Standard psychiatric medications (such as lithium) are anti-suicidal with prolonged use only, and do not impact acute suicidality. A priority for suicide prevention is to define novel treatment targets for safe and rapidly-acting interventions. Recent studies have associated suicide and medically severe suicide attempt (MSSA) with dysregulation of the brain kynurenine pathway (KP), which could predispose to excessive NMDAR activation, a molecular target purportedly involved in rapid improvement of suicidality with agents such as ketamine. AV-101 (4-chlorokynurenine, 4-Cl-KYN) is an oral pro-drug that targets KP dysregulation with downstream NMDAR deactivation. Phase-1 testing showed that AV-101 is metabolized to 7-Cl-KYN in 1.5 to 2 hours after intake.

Objective: Before testing possible anti-suicidal properties, biomarkers need to be defined to show that AV-101 engages the NMDAR. The objective of the current study is to define valid and sensitive neurophysiological markers with a dose-response relationship with AV-101 as evidence of NMDAR engagement, as well as study safety and tolerability.

Methods: The investigators will recruit 12 healthy and non-psychiatrically ill OEF/OIF/OND Veterans (age 25-64) who will receive two single doses of AV-101 (720 mg, 1440 mg) and placebo in a randomized, double-blind, crossover design with one week wash-out between conditions. Neurophysiological measures collected at baseline (pre-treatment) and hourly for 5 hours following medication intake are resting state EEG, Mismatch Negativity amplitude, and P50 sensory gating, measures sensitive to modulation of different NMDAR mechanisms. Repeated measures General Linear Models will be used to test dose-response relationships.

ELIGIBILITY:
Inclusion Criteria

* Age 21-64, inclusive
* US military Veteran
* Healthy volunteer.
* Subject and partner are both using at least 1 medically accepted contraception (double barrier) at randomization until 1 month after single dose

Exclusion Criteria

* History of any Axis 1 psychiatric condition
* History of psychosis in first-degree family members
* History of use of psychoactive medication
* Current use of any medication or vitamins except the pill (women)
* History of use of any substances of abuse, except for alcohol, caffeine, and nicotine
* Positive at tests for alcohol and illicit substance at screening and study visits.
* History of epilepsy, head injury, stroke, primary neurological disorder
* Clinically significant abnormal laboratory values, vital signs or ECG placing participants at risk for serious adverse events as determined by the study physician
* Pregnant or nursing
* Serious, unstable illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2019-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marijn Lijffijt, PhD, Principal Investigator — Baylor College of Medicine and the Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This study is in collaboration with industry partner Vistagen Therapeutics, which provides study medication. Protected health information (PHI) and protected personal information (PII) will not be shared with Vistagen. Study outcomes will be shared as publications.

REFERENCES:
- [Result] Murphy N, Ramakrishnan N, Vo-Le B, Vo-Le B, Smith MA, Iqbal T, Swann AC, Mathew SJ, Lijffijt M. A randomized cross-over trial to define neurophysiological correlates of AV-101 N-methyl-D-aspartate receptor blockade in healthy veterans. Neuropsychopharmacology. 2021 Mar;46(4):820-827. doi: 10.1038/s41386-020-00917-z. Epub 2020 Dec 14. PMID 33318635
- [Derived] Murphy N, Lijffijt M, Ramakrishnan N, Vo-Le B, Vo-Le B, Iqbal S, Iqbal T, O'Brien B, Smith MA, Swann AC, Mathew SJ. Does mismatch negativity have utility for NMDA receptor drug development in depression? Braz J Psychiatry. 2022 Jan-Feb;44(1):61-73. doi: 10.1590/1516-4446-2020-1685. PMID 33825765
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33318635/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with eligible if they were between 18 and 64 years old, a US military veteran, and have no history of psychiatric illness.
Pre-assignment Details: This is a randomized cross-over design, meaning that all subjects received all doses. Total recruited was 18, and total randomized was 12. Ten subjects completed all study visits.
Groups:
- Placebo, Then AV-101 720 mg, Then AV-101 1440 mg: Participants first received a single dose of oral placebo. After at least 3 days wash-out participants got a single dose of oral AV-101 720mg (matching placebo capsules). After at least 3 days wash-out participants got a single dose of oral AV-101 1440mg (matching placebo capsules).
- AV-101 720 mg, Then AV-101 1440 mg, Then Placebo: Participants first received a single dose of oral AV-101 720mg (matching placebo capsules). After at least 3 days wash-out participants got a single dose of oral AV-101 1440mg (matching placebo capsules). After at least 3 days wash-out participants got a single dose of oral placebo.
- AV-101 1440 mg, Then Placebo Then, AV-101 720 mg Then: Participants first received a single dose of oral AV-101 1440mg (matching placebo capsules). After at least 3 days wash-out participants got a single dose of oral placebo. After at least 3 days wash-out participants got a single dose of oral AV-101 720mg (matching placebo capsules).
Period: Period 1
Arm/Group | Placebo, Then AV-101 720 mg, Then AV-101 1440 mg | AV-101 720 mg, Then AV-101 1440 mg, Then Placebo | AV-101 1440 mg, Then Placebo Then, AV-101 720 mg Then
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Placebo, Then AV-101 720 mg, Then AV-101 1440 mg | AV-101 720 mg, Then AV-101 1440 mg, Then Placebo | AV-101 1440 mg, Then Placebo Then, AV-101 720 mg Then
Started | 4 | 4 | 4
Completed | 3 | 4 | 3
Not Completed | 1 | 0 | 1
Not completed — Did not receive treatment due to loss of contact | 1 | 0 | 1
Period: Period 3
Arm/Group | Placebo, Then AV-101 720 mg, Then AV-101 1440 mg | AV-101 720 mg, Then AV-101 1440 mg, Then Placebo | AV-101 1440 mg, Then Placebo Then, AV-101 720 mg Then
Started | 3 | 4 | 3
Completed | 3 | 4 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Twelve subjects started the study; 10 completed all visits. Baseline outcomes are provided for the 12 subjects who started the study.
Groups:
- All Study Participants: All 12 study participants who started the study
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.33 (6.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity (self-report)
  Participants
    Hispanic or Latino | 7
    Not Hispanic or Latino | 5
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race (self-report)
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 10
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean 40-Hz Auditory Steady State Response Power
Description: Mean power (in microVolt squared; uV^2) of 40-Hz Auditory Steady State Response (ASSR; an auditory task using 40Hz click trains) calculated across 38-42Hz.
  Mean +/- SE across pre-treatment baseline and 4 post-treatment measures one every hour controlled for time, with outcomes the mean per treatment arm obtained from Linear Mixed Model analysis.
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: uV^2
Groups:
- Placebo: Placebo
  Placebo: Single dose of 4 placebo oral capsules
- AV-101 720 mg: One time 720 mg L-4-Chlorokynurenine
  AV-101 720 mg: Single dose of 2 360 mg AV-101 oral capsules + 2 placebo oral capsules
- AV-101 1440 mg: One time 1440 mg L-4-Chlorokynurenine
  AV-101 1440 mg: Single dose of 4 360 mg AV-101 oral capsules
Arm/Group | Placebo | AV-101 720 mg | AV-101 1440 mg
Number analyzed (Participants) | 10 | 10 | 10
uV^2 | 0.34 (0.11) | 0.43 (0.11) | 0.60 (0.11)

2. Secondary Outcome: Peak Change in Plasma Concentration of AV-101 Marker 4-Chloro-kynurenine
Description: Assesses the peak change from baseline and corrected for placebo (placebo set at 0) across a 4 hours time frame after drug intake. 4-Chloro-kynurenine is the main ingredient of AV-101 and is a precursor of 7-Chloro-kynurenic acid.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: ng/Ml
Groups:
- Placebo: Outcomes across placebo
- AV-101 720 mg: Outcomes across AV-101 720mg
- AV-101 1440 mg: Outcomes across AV-101 1440mg
Arm/Group | Placebo | AV-101 720 mg | AV-101 1440 mg
Number analyzed (Participants) | 10 | 10 | 10
ng/Ml | 0 (0) | 28,532 (21,462) | 51,450 (21,182)

3. Secondary Outcome: Peak Change in Plasma Concentration of AV-101 Marker 7-Chloro-kynurenic Acid
Description: Assesses the peak change from baseline and corrected for placebo (placebo set at 0) across a 4 hours time frame after drug intake. 7-Chloro-kynurenic acid is the main metabolite of AV-101 (4-Chloro-kynurenine).
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: ng/Ml
Arm/Group | Placebo | AV-101 720 mg | AV-101 1440 mg
Number analyzed (Participants) | 10 | 10 | 10
ng/Ml | 0 (0) | 93 (48) | 412 (473)

4. Secondary Outcome: Mean Systolic Blood Pressure
Description: Systolic blood pressure Mean +/- SE averaged across all timepoints (including baseline). Systolic blood pressure was measured 15 minutes before drug intake and every 15 minutes from drug intake until 5 hours after intake controlled for time, with outcomes the mean per treatment arm obtained from Linear Mixed Model analysis.
Time Frame: 5 hours
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | AV-101 720 mg | AV-101 1440 mg
Number analyzed (Participants) | 10 | 10 | 10
mm Hg | 122.5 (2.7) | 119.6 (2.7) | 120.1 (2.7)

5. Secondary Outcome: Mean Diastolic Blood Pressure
Description: Diastolic blood pressure Mean +/- SE averaged across all timepoints (including baseline). Diastolic blood pressure was measured 15 minutes before drug intake and every 15 minutes from drug intake until 5 hours after intake controlled for time, with outcomes the mean per treatment arm obtained from Linear Mixed Model analysis
Time Frame: 5 hours
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | AV-101 720 mg | AV-101 1440 mg
Number analyzed (Participants) | 10 | 10 | 10
mm Hg | 80.8 (2.35) | 79 (2.35) | 76.3 (2.35)

6. Secondary Outcome: Mean Pulse
Description: Pulse Mean +/- SE averaged across all timepoints (including baseline). Pulse was measured 15 minutes before drug intake and every 15 minutes from drug intake until 5 hours after intake controlled for time, with outcomes the mean per treatment arm obtained from Linear Mixed Model analysis
Time Frame: 5 hours
Measure: Mean (Standard Error); unit: beat per minute (bpm)
Arm/Group | Placebo | AV-101 720 mg | AV-101 1440 mg
Number analyzed (Participants) | 10 | 10 | 10
beat per minute (bpm) | 68.8 (1.82) | 70.5 (1.82) | 69.9 (1.82)

7. Secondary Outcome: Mean Profile of Moods Scale Total Score
Description: POMS total score Mean +/- SE averaged across all timepoints (including baseline). Systolic blood pressure was measured directly before drug intake and every hours from drug intake until 5 hours after intake controlled for time, with outcomes the mean per treatment arm obtained from Linear Mixed Model analysis
  The POMS is a 40 item scale. Each item is scored on a 0 (absent) - 4 (extreme) scale. POMS total score ranges from 0 to 160. Higher scores mean more extreme dysregulated mood. Subscales are tension (6 items; score anger 0-24), depression (6 items, range 0-24), fatigue (5 items, range 0-20), vigor (6 items, range 0-24), confusion (5 items, range 0-20), anger (7 items, range 0-28), and mania-related affect (5 items, range 0-20).
Time Frame: 5 hours
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | AV-101 720 mg | AV-101 1440 mg
Number analyzed (Participants) | 10 | 10 | 10
Units on a scale | 11.6 (1.65) | 12 (1.65) | 11.6 (1.65)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Asked by study team if experiencing any health complications last 24 hours since study intake. Any health complications not related to the study medication were also asked about when subjects at study visits from the moment that they were enrolled in the study until they had completed the study.
Arm/Group | Placebo | AV-101 720 mg | AV-101 1440 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | AV-101 720 mg (N=12) | AV-101 1440 mg (N=12)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — diarrhea
Elation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Elation (self-report)

LIMITATIONS AND CAVEATS:
The small number of subjects limits power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT03583554/Prot_000.pdf